CLINICAL TRIAL: NCT02714647
Title: The Role of an Attention Demanding Activity for Priming Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Walter, Graduate Student, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 82401
Record Dates: First submitted 2016-03-02; First posted 2016-03-21 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Basic Motor Learning Problem
Keywords: motor learning; attention; priming; rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): This group will perform the attention demanding activity (a variant of the Simon Task) with a focus on accuracy over speed prior to practicing the motor task. Participants will also have extended deadlines (750 ms) throughout the task to ensure an accuracy preference. Participants will then perform 50 trials of the simulated feeding task where they will spoon two raw kidney beans at a time from a center proximal "start" cup to three distal "target" cups positioned 16 cm away at 45°, 90°, and 135° around the start cup as fast as possible using the non-dominant hand. Spooning two beans between the start cup and a target cup is considered one repetition where each trial will consist of 15 repetitions.
  Interventions: Behavioral: Attentional prime
- Control (Sham Comparator): This group will perform the attention demanding activity (a variant of the Simon Task) with a focus on speed over accuracy prior to practicing the motor task. Participants will also have short deadlines (250 ms) throughout the task to ensure a speed preference. Participants will then perform 50 trials of the simulated feeding task where they will spoon two raw kidney beans at a time from a center proximal "start" cup to three distal "target" cups positioned 16 cm away at 45°, 90°, and 135° around the start cup as fast as possible using the non-dominant hand. Spooning two beans between the start cup and a target cup is considered one repetition where each trial will consist of 15 repetitions.
  Interventions: Behavioral: Sham prime

INTERVENTIONS:
Behavioral: Attentional prime
  Arms: Experimental
Behavioral: Sham prime
  Arms: Control

SUMMARY:
The purpose of this study is to determine if priming attention prior to practicing a motor task will have an effect on the ability to acquire and learn that motor task. The investigators hypothesize that the acquisition and learning of a motor task will improve if attention is primed prior to practicing that motor task when compared to a group who does not receive the prime.

DETAILED DESCRIPTION:
This proposed study is a randomized trial on the effects of using an attention demanding prime prior to practicing a previously untrained motor task in a population of young and healthy individuals. Therefore, The investigators will randomize a group into a motor learning paradigm. The experimental group will prime with an activity that requires high attention demands . The control group will perform an activity that is matched for practice amount but requires less attention demands. Both groups will perform this activity immediately prior to practicing a previously untrained motor task. The objectives of our aims will be to compare the experimental group to the control group to determine the effects of the attention demanding prime on the amount, rate, and transfer of acquisition and learning of the motor task.

On day one of the study, participants will be consented. Demographic information, participant's hand dominance (self-report), and level of arousal will then be documented. Level of arousal will be assessed by using the Stanford Sleepiness Scale. Each participant will then perform baseline measures on the previously untrained motor task, a functional task that simulates feeding, and two other motor task that will not be practiced which will be used to determine transfer of the practiced task. One task will be a card sorting task, which shares similar spatio-temporal characteristics to the simulated feeding task. The other transfer task will be a buttoning task which has dissimilar spatio-temporal characteristics when compared to the simulated feeding task. Baseline measurements will consists of two trials for each motor task and trial order will be randomized between all tasks. Each participant will then be randomized into either the experimental group or the control group using a block randomization technique. Participants randomized to the experimental group will perform the attention demanding task, a variant of the Simon Task, and will be told to emphasize accuracy over speed in order to prime for attention. Participants randomized to the control group will perform a similar task; however will be told to emphasize speed over accuracy; thereby creating a sham prime. Following completion of the cognitive tasks, both groups will immediately begin practicing 50 trials of the simulated feeding task. Following completion of practice on the simulated feeding task, participants will again perform 2 trials of both the card sorting task and the buttoning task to determine transfer of the unpracticed task. Participants will then return on day 2 and will perform 2 trials of the simulated feeding task to assess for short term retention. Participants will again return on day 8 and will complete two trials of each motor task (simulated feeding task, card sorting task, and buttoning task) to determine delayed retention and transfer.

The Attention Demanding Activity: The attention demanding activity will be a variant of the Simon Task, a choice reaction time task. In this task, participants will be instructed to respond as quickly and accurately as possible, pushing one of two buttons corresponding to the direction of arrows presented visually on a computer screen, ignoring the spatial location of the arrows. Arrows will be presented in one of two conditions: congruent and incongruent. Each arrow will be preceded by a fixation cross presented for 250 milliseconds in the center of the display followed by a blank screen for 100 milliseconds. The arrow will then be presented until the participant responds or 250 milliseconds or 750 milliseconds elapse depending on the group. In the congruent conditions, arrows will appear on the same side of the space as the direction they are facing (e.g. a right facing arrow on the right side of the space). In the incongruent condition, arrows will be presented on the opposite side of the space as the direction they are facing (e.g. a right facing arrow on the left side of the space). There will be a high proportion of congruent trials (75%; 480 trials) to incongruent trials (25%; 160 trials). In addition to verbal instructions, response deadlines will be in place. In order to ensure that the experimental group focuses on accuracy over speed, the deadlines throughout their activity will be 750 milliseconds. The control group will only have 250 milliseconds to respond to the on-screen stimulus which will ensure a focus on speed over accuracy. If a deadline is not met on a given trial, a message will appear to the participant as "Deadline Missed. Faster!" Every 15 trials, this was evaluated, and if more than 33% of deadlines are missed, a message will appear indicating that the participants are missing too many deadlines and that it is imperative that the deadlines be met, even if errors result.

The previously untrained motor task: The investigators have chosen to use a functional upper extremity motor task that simulates feeding. This task requires participants to spoon beans (kidney, raw) from a central, proximal "start" cup to 3 distal "target" cups as fast as possible. The cups (9.5 centimeters in diameter) will be secured to a board with 3 cups secured radially at 45 degrees, 90 degrees, and 135 degrees around the start cup at a distance of 16 centimeters. The start cup will be oriented along the participant's midline and 15 centimeters in front of the seated participant. One repetition of the motor task will consist of spooning 2 beans at once from the start cup to a target cup with the non-dominant hand, with one trial equaling 15 repetitions. During each trial, participants will move first to the ipsilateral target cup, next to the center target cup, and then to the contralateral cup, relative to the hand used (right vs. left). This sequence will be repeated five times to complete the trial. The participant will begin each trial with their non-dominant hand to the side of the spoon. Each trial will begin as the administrator gives a verbal cue "go" and will end when the spoon is returned to the starting position (5 centimeters lateral to the start cup). The time it takes to complete the 15 repetitions ("trial time") will be the measure of performance, with faster times indicating better performance. All trials will be timed to the nearest 100th of a second via stopwatch. Participants will be given no explicit feedback (i.e. knowledge of performance or results) after each trial. They will also not be encouraged or coached to use a specific pattern of upper extremity kinematics during training.

Transfer task that has similar spatio-temporal characteristics: This task will be a card sorting task. This task requires participants to place a standard playing card from a central, proximal "start" box to three distal target boxes as fast as possible. The boxes (9 centimeters X 9 centimeters) will be secured to a board with 3 boxes secured radially at 45 degrees, 90 degrees, and 135 degrees around the start box at a distance of 16 centimeters. The start box will be oriented along the participant's midline and 15 centimeters in front of the seated participant with the cards face down. One repetition of the motor task will consist of placing one card at a time; face up, from the start box to a target box with the non-dominant hand with one trial equaling 15 repetitions. During each trial, participants will move first to the ipsilateral target box, next to the center target box, and then to the contralateral box, relative to the hand used (right vs. left). This sequence will be repeated ten times to complete the trial. The participant will begin each trial with their non-dominant hand to the side of the start box. Each trial will begin as the administrator gives a verbal cue "go" and will end when the participant places their hand back at the starting location after the last card is at rest in the target box. The time it takes to complete the 30 repetitions ("trial time") will be the measure of performance, with faster times indicating better performance. All trials will be timed to the nearest 100th of a second via stopwatch. Participants will be given no explicit feedback (i.e. knowledge of performance or results) after each trial. They will also not be encouraged or coached to use a specific pattern of upper extremity kinematics during training.

Transfer task that has dissimilar spatio-temporal characteristics: This task will require fastening buttons sequentially. At the start of each trial, participants will begin buttoning the top of ten buttons (3 centimeters apart) that will be sewed 2 centimeters apart vertically on a piece of plain weave cotton fabric. Both pieces of the fabric will be secured to a wooden board with the placket centered in line with the subject's non-dominant shoulder. The button side of the fabric will be folded onto the board, while the buttonhole side of the fabric will be unfolded onto the table prior to each trial. Buttons will be fastened through horizontal buttonholes in a left over right order, relative to the participant. Participants will fasten all ten buttons sequentially and then will unfasten each button in the reverse order using their non-dominant hand. The time it takes to fasten and unfasten all 10 buttons will be the trial time or measure of performance, with faster times indicating better performance. All trials will be timed to the nearest 100th of a second via stopwatch. Participants will be given no explicit feedback (i.e. knowledge of performance or results) after each trial. They will also not be encouraged or coached to use a specific pattern of upper extremity kinematics during training. This task will be performed with the subject's non-dominate upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35

Exclusion Criteria:

* Present with acute medical problems or orthopedic injuries that would limit participation in the motor task
* Uncorrected vision loss
* Has a neurological disease
* Consider themselves ambidextrous

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-26 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance time (trial time) on the simulated feeding task at the end of training | Day one
  Average trial time on the simulated feeding task at the end of training compared to trial time on the simulated feeding task at baseline.
Change from baseline performance time (trial time) on the simulated feeding task at one-day retention | Day two
  Average trial time of two trials on the simulated feeding task on day two compared to trial time on the simulated feeding task at baseline.
Change from baseline performance time (trial time) on the simulated feeding task at eight-day retention | Day eight
  Average trial time of two trials on the simulated feeding task on day eight compared to trial time on the simulated feeding task at baseline.

SECONDARY OUTCOMES:
Change from baseline in performance time (trial time) on the untrained similar transfer task (card sorting task) at the end of training | Day one
  Average trial time on the card sorting task after training on the simulated feeding task compared to trial time on the card sorting task at baseline.
Change from baseline in performance time (trial time) on the untrained similar transfer task (card sorting task) at day eight | Day eight
  Average trial time on the card sorting task performed on day eight compared to trial time on the card sorting task at baseline.
Change from baseline in performance time (trial time) on the untrained dissimilar transfer task (buttoning task) at the end of training | Day one
  Average trial time on the buttoning task after training on the simulated feeding task compared to trial time on the buttoning task at baseline.
Change from baseline in performance time (trial time) on the untrained dissimilar transfer task (buttoning task) at day eight | Day eight
  Average trial time on the buttoning task performed on day eight compared to trial time on the buttoning task at baseline.
Rate of improvement | trial time (in seconds) during practice (day 1) will be plotted as a function of trial number (1-50)
  Rate of improvement (c) will be modeled using an exponential decay function: y=a + be (exp[-x/c]), where a is the final trial time value that the exponential decay function approaches (i.e. asymptote), b is the scale of the learning from the first trial time to the value a, x is the trial number, 1/c is the number of trials needed to obtain asymptote (i.e. 1-e-1).
Priming measures | when performed during the priming/sham priming activities on day one
  accuracy (% correct) and reaction time ( in ms). This will allow us to ensure that the participant's have completed the task according to the directions.
Level of arousal | Day one
  using the Stanford Sleepiness Scale to ensure that the motor improvement is not due to level of arousal.
Level of arousal | Day two
  using the Stanford Sleepiness Scale to ensure that the motor improvement is not due to level of arousal.
Level of arousal | Day eight
  using the Stanford Sleepiness Scale to ensure that the motor improvement is not due to level of arousal.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah College of Health; Division of Occupational Therapy, Salt Lake City, Utah, United States